CLINICAL TRIAL: NCT06651125
Title: EXPLORING the IMPACT of SUPERVISED PHYSICAL ACTIVITY INTERVENTION on CACHECTIC CANCER PATIENTS: a PRELIMINARY STUDY
Acronym: APACAVIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rennes 2 (Other)
Responsible Party: Principal Investigator, Peyrachon Romane, MD, University of Rennes 2
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APACAVIR
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Cancer Cachexia
Keywords: Cancer Cachexia; Exercise; Adapted Physical Activity; Resistance training; Endurance training; Body composition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cachectic Cancer Patients (Experimental)
  Interventions: Other: Adapted Physical Activity

INTERVENTIONS:
Other: Adapted Physical Activity — Patients in the Adapted Physical Activity arm realized a 12-weeks supervised exercise program. The supervised PA intervention consisted of two sessions per week. Each session lasted one hour and was divided into 30 minutes of aerobic exercise using an ergometer (treadmill and/or bicycle), followed by 30 minutes of resistance exercises involving major muscle groups, with or without small equipment such as dumbbells, resistance bands, and balls. The exercise regimen was carried out at an intensity ranging from 50% to 70% of the heart rate reserve, with a rate of perceived exertion (RPE) set at 4 on a Borg scale of 0 to 10. A total of 24 sessions were planned. There was also the option to incorporate a 45-minute session of moderate-intensity water aerobics into the weekly routine.

SUMMARY:
The goal of this project is to observe the benefits induced by physical activity during a supervised adapted physical activity program at SPORMED.

Methodology: By agreeing to participate in this study, participation in a supervised adapted physical activity (APA) program at SPORMED and undergoing a series of evaluations will be required.

At the start of the adapted physical activity program (T0), two APA sessions per week will be carried out for eight weeks. These group sessions, involving four participants, last 1 hour and are divided into 30 minutes of aerobic work on an ergometer followed by 30 minutes of muscle strengthening of the four limbs and core exercises, with or without small equipment. There is also the option to add a 45-minute balneotherapy session once a week, if desired and no contraindications are present. At the end of the eight weeks (T1), a follow-up phase begins, consisting of one APA session per week for another eight weeks. The session will be identical to the previously described sessions and can also be complemented by a balneotherapy session. The APA program will conclude after these 12 weeks (T2). A total of 24 indoor sessions will be offered, which can be supplemented by 12 balneotherapy sessions. Attendance at the sessions will be recorded.

Additionally, a series of evaluations will take place at T0, T1, and T2. These include physical and anthropometric assessments at SPORMED lasting approximately 30 minutes. They involve weight and body composition evaluation (2 minutes), height measurement (1 minute), waist and hip circumference measurements using a tape measure (2 minutes). Next, an upper limb strength test will be conducted, involving three maximal contractions during a handgrip test with 30-second rest intervals (2 minutes), followed by a lower limb strength test, which involves performing as many sit-to-stand repetitions from a chair with a backrest and without armrests as possible in 30 seconds (30 seconds). Then, a balance test, including bipodal and unipodal stance (30 seconds on both feet, followed by each foot individually), will be performed, and finally, a 6-minute walking test, during which the longest possible distance must be covered (without running) in 6 minutes (6 minutes, with the option to stop if necessary).

Additionally, four self-assessment questionnaires on quality of life, fatigue, physical activity level, and food consumption must be completed at home (about 20 to 30 minutes).

DETAILED DESCRIPTION:
Patient volunteers were referred to Spormed sports medicine center by an oncologist and/or general practitioner. To be eligible for the study, participants had to be over 18 years old and have a diagnosis of cachexia-inducing cancer. Metastasis could be present or not. Participants could either be undergoing treatment or have completed treatment within the last year. They had to be able to participate in physical activity (PA). Additionally, registration with the French health insurance system and having French as the primary language were required. Those who could not report weight changes in the last 6 months, individuals with disabilities preventing them from understanding study instructions, and those with medical contraindications for PA were excluded from the study.

Participants were assigned to the "cachectic" group if classified in categories 3 or 4 of the Martin and colleagues classification. This classification is based on two criteria: percentage of weight loss in the past six months and body mass index. Participants classified as grades 0, 1, or 2 were included in the "non-cachectic" group. The "non-cachectic" group was matched to the "cachectic" group based on sex, age, and number of PA sessions completed. The aim was to verify whether the recognized effects of APA in non-cachectic individuals could be transferred to cachectic participants, with matching on the compliance variable to avoid an effect related to the amount of practice. Matching tumor type was not possible, as certain tumors are almost exclusively cachectizing.

Supervised Physical Activity Intervention:

The supervised PA intervention consisted of two sessions per week over a span of 12 weeks. Each session lasted one hour and was divided into 30 minutes of aerobic exercise using an ergometer (treadmill and/or bicycle), followed by 30 minutes of resistance exercises involving major muscle groups, with or without small equipment such as dumbbells, resistance bands, and balls. The exercise regimen was carried out at an intensity ranging from 50% to 70% of the heart rate reserve, with a rate of perceived exertion (RPE) set at 4 on a Borg scale of 0 to 10. A total of 24 sessions were planned. There was also the option to incorporate a 45-minute session of moderate-intensity water aerobics into the weekly routine.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Diagnosis of cancer cachexia
* Able to participate in exercise program
* Registered with the French health insurance system
* Understanding and speaking French

Exclusion Criteria:

* Medical contraindications for exercise
* No report of weight changes in the last 6 months
* Disabilities to understand the study instructions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Attrition rate | Through study completion, an average of 3 months
  Attrition rate was the number of patients who completed the baseline and follow-up assessments versus the number of patients who completed initial assessments and started the program
Compliance rate | Through study completion, an average of 3 months
  Compliance rate was the number of sessions completed out of the number of sessions prescribed
Serious adverse events | Through study completion, an average of 3 months
  Serious adverse events occurring during the exercise program

SECONDARY OUTCOMES:
Nutritional status | Through study completion, an average of 3 months
  Food intake was evaluated using the analog scale Simple Evaluation of Food Intake (SEFI®)
Body weight | Through study completion, an average of 3 months
  Body weight (kg)
Fat mass | Through study completion, an average of 3 months
  Fat mass was assessed using bioelectrical impedance analysis
Lean mass | Through study completion, an average of 3 months
  Lean mass (kg) was assessed using bioelectrical impedance analysis (Tanita, DC-360).
Physical activity level | Through study completion, an average of 3 months
  PA level was assessed using the International Physical Activity questionnaire Short-Form (IPAQ-SF). This 7 items questionnaire covers overall PA, broken down into intense, moderate and walking activities, and the level of sedentary lifestyle over the past seven days.
Functional aerobic capacity | Through study completion, an average of 3 months
  Functional aerobic capacity was measured using the 6-minute walk test. Patients were instructed to walk back and forth along a 20-meter corridor to cover the greatest distance at constant speed. After 6 minutes, the distance walked was recorded in meters.
Lower limb strength | Through study completion, an average of 3 months
  Proximal lower limb strength was evaluated using a 30-second (sec) chair sit-to-stand test. Patients were instructed to rise from a seated position to a standing position and return to seating, without assistance and without using their arms, as many times as possible within 30 sec. The number of complete stands within this period was recorded.
Grip strength | Through study completion, an average of 3 months
  Grip strength was measured using a Hand Grip Digital Dynamometer (Takei 5401 Hand Grip Digital Dynamometer). The test was performed with patients in a sitting position, with both feet touching the ground, hand holding the dynamometer, elbow flexed at 90° and shoulder adducted. The participant were instructed to squeeze the handle with maximum force for 3 sec. The test was repeated three times, with 30 seconds of recovery time between each effort. The highest value of the three repetition was retained in kilograms (kg) for each hand.
Balance ability | Through study completion, an average of 3 months
  Static balance ability was evaluated using the single-leg stance test. The time the patient-maintained balance on one leg with eyes open was recorded (maximum 30 sec).
Perceived Fatigue | Through study completion, an average of 3 months
  Fatigue was assessed using the Multidimensional Fatigue Inventory (MFI). The questionnaire comprises 20 statements in which the patient positions himself on a Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree").

CONTACTS AND LOCATIONS:
Locations (1):
- SPORMED, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No